CLINICAL TRIAL: NCT01169207
Title: Johns Hopkins Crohn's Disease and Ulcerative Colitis Study
Status: Active, not recruiting | Type: Observational
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Other Study IDs: NA_00041583
Record Dates: First submitted 2010-07-23; First posted 2010-07-26 (Estimated); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Inflammatory Bowel Disease
Keywords: Inflammatory Bowel Disease; Crohn's Disease; Ulcerative Colitis; Indeterminate Colitis; IBD; CD; UC; IC
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood and derivative from blood, saliva
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Unaffected: Individuals who do not have IBD
- Affected: Individuals with IBD

SUMMARY:
Inflammatory bowel disease (IBD), including Crohn's disease (CD) and ulcerative colitis (UC), is a idiopathic, chronic and frequently disabling inflammatory disorder of the intestines characterized by a dysregulated mucosal immune response that affect more than a million Americans. This current protocol was established in 1996 with the goal of identifying the genetic and environmental components that contribute to the development of IBD, especially in families.

DETAILED DESCRIPTION:
The investigators initiated this research study in 1996 with the overall goal of identifying IBD susceptibility genes. In the beginning, the major focus was recruitment of multiply affected IBD pedigrees for linkage studies, but the investigators have since expanded the study to include singleton cases and spousal/friend as well as population controls for comparison purposes The investigator's recruitment goal is 2500 subjects.

Blood samples obtained from participants are used to isolate lymphocytes for storage, serum for serological analysis of antibodies and other proteins relevant to IBD and DNA for genotyping or sequencing. Lymphocytes may be transformed with EBV to establish immortalized lymphoblastoid cell lines. These cell lines can be used as a secondary DNA source or to study IBD relevant gene, protein expression and cell function

ELIGIBILITY:
Inclusion Criteria:

ADULTS:

* Patients with IBD and family members who have or do not have IBD.
* People that do not have IBD nor have a family member with IBD needed for comparison purposes.

CHILDREN:

* Children age 5 or older with IBD and family members who have or do not have IBD.
* Children that do not have IBD nor have a family member with IBD needed for comparison purposes.

Exclusion Criteria:

* The only exclusions are age parameters and health reasons that would preclude enrollment; such as, for anemic patients. Blood-draws on anemic patients may, in certain medical cases, pose a health risk; therefore, the investigators request that if the participants are anemic that the participants present a letter from the participant's personal physician giving explicit permission for the participant to join if at the time it is clinically advisable.

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: IBD patients are primarily recruited at the Johns Hopkins inpatient and outpatient units. However, individuals may contact by phone, mail or email after hearing about the study.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 1996-07; Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Genetics of IBD | Single visit, approximately 1 hour

CONTACTS AND LOCATIONS:
Overall Officials: Florin Selaru, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University, Baltimore, Maryland, United States